CLINICAL TRIAL: NCT03212365
Title: Minimization of Bleeding Related Adverse Drug Events in Plastic & Reconstructive Surgery Patients Randomized to Different Postoperative Anticoagulant Regimens
Brief Title: Minimization of Bleeding Related Adverse Drug Events in Plastic & Reconstructive Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Stanford University (Other)
Responsible Party: Principal Investigator, Christopher Pannucci, Assistant Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 100416
Record Dates: First submitted 2017-07-06; First posted 2017-07-11 (Actual); Results first posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-08

CONDITIONS: Venous Thromboembolism; Deep Venous Thrombosis; Pulmonary Embolus; Reconstructive Surgery
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis; Pulmonary Embolism

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into one of two groups (enoxaparin 40mg twice daily or enoxaparin 0.5mg/kg twice daily, rounded to the nearest milligram).
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fixed Dose (Other): Participants will receive 40 mg enoxaparin twice daily
  Interventions: Drug: Fixed dose
- Variable Dose (Experimental): Participants will receive 0.5mg/kg enoxaparin twice daily
  Interventions: Drug: Variable dose

INTERVENTIONS:
Drug: Fixed dose — Participants will receive 40 mg enoxaparin twice daily
  Arms: Fixed Dose
Drug: Variable dose — Participants will receive 0.5mg/kg enoxaparin twice daily
  Arms: Variable Dose

SUMMARY:
Plastic and reconstructive surgeons consistently create large, raw surfaces as part of their operative procedures. Thus, plastic & reconstructive surgery patients are among those at highest risk for anticoagulant-associated bleeding adverse drug events (ADEs). This study seeks to optimize both the safety and effectiveness of post-operative enoxaparin by comparing aFXa levels, bleeding events, and VTE events among plastic & reconstructive surgery patients randomized to receive two different enoxaparin dose regimens.

DETAILED DESCRIPTION:
Plastic and reconstructive surgeons consistently create large, raw surfaces as part of their operative procedures. Thus, plastic & reconstructive surgery patients are among those at highest risk for anticoagulant-associated bleeding adverse drug events (ADEs). Our preliminary data has shown that a fixed, or "one size fits all" dose of enoxaparin, an anticoagulant, can allow a high proportion of patients to have appropriately thinned blood, measured by anti-Factor Xa (aFXa) levels. Patients with adequate aFXa levels are known to have significantly decreased venous thromboembolism risk (VTE), which is desirable. However, 30% of patients who receive fixed dose enoxaparin have blood that is too thin. Patients who are over-anticoagulated are significantly more likely to have ADEs including bleeding requiring return to the operating room, need for blood transfusion, or death. The optimal way to dose enoxaparin to minimize ADEs remains unknown. This study seeks to optimize both the safety and effectiveness of post-operative enoxaparin by comparing aFXa levels, bleeding events, and VTE events among plastic & reconstructive surgery patients randomized to receive two different enoxaparin dose regimens.

ELIGIBILITY:
Inclusion Criteria:

* receiving plastic and reconstructive surgery under general anesthesis
* Expected post-operative stay of 2 days or more

Exclusion Criteria:

* Contraindication to use of enoxaparin
* intracranial bleeding/stroke
* Hematoma or bleeding disorder
* Heparin-induced thrmbocytopenia positive
* Creatinine clearance less than or equal to 30 mL/min
* Serum creatinine greater than 1.6 mg/dL
* epidural anesthesia
* patients placed on non-enoxaparin chemoprophylaxis regimens
* gross weight exceeding 150kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 295 (Actual)
Dates: Start 2017-07-03 (Actual); Primary Completion 2019-06-02 (Actual); Study Completion 2019-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Puccini, MD, Principal Investigator — University of Utah
Locations (2):
- United States (2):
  - Stanford University, Stanford, California
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Derived] Pannucci CJ, Fleming KI, Varghese TK Jr, Stringham J, Huang LC, Pickron TB, Prazak AM, Bertolaccini C, Momeni A. Low Anti-Factor Xa Level Predicts 90-Day Symptomatic Venous Thromboembolism in Surgical Patients Receiving Enoxaparin Prophylaxis: A Pooled Analysis of Eight Clinical Trials. Ann Surg. 2022 Dec 1;276(6):e682-e690. doi: 10.1097/SLA.0000000000004589. Epub 2020 Oct 19. PMID 33086312

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fixed Dose | Variable Dose
Started | 151 | 144
Completed | 128 | 130
Not Completed | 23 | 14
Not completed — Discharged prior to Xa level | 12 | 8
Not completed — Bled requiring enoxaparin cessation | 4 | 2
Not completed — Refused study medication | 3 | 0
Not completed — Initiated heparin infusion on floor | 1 | 1
Not completed — Unexpected return to OR | 1 | 1
Not completed — Medication distribution error | 1 | 0
Not completed — Required epidural placement | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — developed acute renal failure | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fixed Dose | Variable Dose | Total
Number analyzed (Participants) | 151 | 144 | 295
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.0 (15.6) | 52.7 (14.8) | 50.8 (15.3)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 81 | 70 | 151
  Male | 70 | 74 | 144
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 137 | 135 | 272
  African American | 1 | 0 | 1
  Native American/Alaskan Native | 1 | 0 | 1
  Hispanic or Latino | 11 | 8 | 19
  Pacific Islander | 1 | 0 | 1
  Other | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 151 | 144 | 295

OUTCOME MEASURES:

1. Primary Outcome: Avoidance of Under-anticoagulation (Peak aFXa <0.2 IU/mL)
Description: Avoidance of under-anticoagulation (peak aFXa <0.2 IU/mL)
Time Frame: Four hours following third enoxaparin dose
Measure: Number; unit: percentage of participants
Arm/Group | Fixed Dose | Variable Dose
Number analyzed (Participants) | 128 | 130
percentage of participants | 76.6 | 79.9

2. Primary Outcome: Avoidance of Over-anticoagulation (Peak aFXa >0.4 IU/mL)
Description: Avoidance of over-anticoagulation (peak aFXa >0.4 IU/mL)
Time Frame: Four hours following third enoxaparin dose
Measure: Number; unit: percentage of participants
Arm/Group | Fixed Dose | Variable Dose
Number analyzed (Participants) | 128 | 130
percentage of participants | 82.2 | 90.6

3. Secondary Outcome: Percentage of Participants With Venous Thromboembolism Events
Description: Any symptomatic venous thromboembolism events, including deep venous thrombosis or pulmonary embolus occurring within 90 days of surgery
Time Frame: 90 days
Measure: Number; unit: percentage of patients
Arm/Group | Fixed Dose | Variable Dose
Number analyzed (Participants) | 151 | 144
percentage of patients | 0.66 | 0.69

4. Secondary Outcome: Percentage of Patients With Bleeding Events
Description: Bleeding events requiring alteration in the course of care within 90 days of surgery
Time Frame: 90 days
Measure: Number; unit: percentage of patients
Arm/Group | Fixed Dose | Variable Dose
Number analyzed (Participants) | 151 | 144
percentage of patients | 6.0 | 8.3

ADVERSE EVENTS:
Time Frame: 90 days
Description: Study team performed chart review and made mandatory phone contact with patients at 90 days to identify adverse events.
Arm/Group | Fixed Dose | Variable Dose
All-Cause Mortality (participants affected / at risk) | 1/151 | 0/144
Serious Adverse Events (participants affected / at risk) | 0/151 | 0/144
Other Adverse Events (participants affected / at risk) | 0/151 | 0/144

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-06): https://cdn.clinicaltrials.gov/large-docs/65/NCT03212365/Prot_SAP_000.pdf